CLINICAL TRIAL: NCT01293825
Title: Ziprasidone Switching in Response to Adherence and Psychotropic-Related Weight Gain Concerns Among Patients With Bipolar Disorder
Brief Title: Ziprasidone Switching in Response to Adherence and Psychotropic-Related Weight Gain Concerns Among Patients With Bipolar Disorder (Zip Ad)
Acronym: Zip Ad
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Martha Sajatovic, Professor of Psychiatry, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pfizer IIR-WS883414
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2014-04-22 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Medication Adherence; Bipolar Disorder
MeSH Terms: conditions — Medication Adherence; Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Medication Adherence Bipolar Disorder (Experimental): There was only one group in this study. All participants received the study drug Ziprasidone.
  Interventions: Drug: ziprasidone

INTERVENTIONS:
Drug: ziprasidone — Patients will identify which psychotropic they currently receive that causes the most weight-gain concern. For individuals on multiple drugs, one drug must be identified as the "offending agent". Study psychiatrist will switch the "offending agent" to ziprasidone. Participants will be switched to ziprasidone per package insert. Patients will be maintained on ziprasidone for 12 weeks (active part of study). After the active part of the study they will return to the care of their normal clinical provider who will determine whether they will continue on ziprasidone.
  Other Names: Geodon

SUMMARY:
Psychotropic-related weight gain is a common concern among patients with bipolar disorder (BD). This concern affects an individual's satisfaction with treatment and may lead to reduced adherence and illness relapse. Patient-focused care is attentive to patient concerns while at the same time utilizing evidence-based treatments. Ziprasidone is currently FDA approved for the maintenance treatment of BD. Ziprasidone may be associated with less weight gain compared to some alternative BD maintenance treatments. The proposed project will evaluate how switching to ziprasidone may affect patient adherence, drug attitudes, satisfaction with care and clinical outcomes (psychiatric symptoms, functional status, weight) among BD patients concerned with weight gain.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Type I or II BD for at least 6 months (confirmed with MINI)
2. On maintenance evidence-based treatment for BD (lithium, antipsychotic, anticonvulsant)
3. Have weight gain concerns that individual believes are related to BD medication treatment
4. Sub-optimal adherence as measured by the Tablet Routines Questionnaire (TRQ) and which the patient feels is related to weight gain concerns. TRQ threshold will be defined as missing an average of 20% or more of all prescribed BD treatment in the last week or month or missing 20% or more of the "offending agent" in the last week or last month. This is consistent with methodologies in PIs previous BD adherence studies

Exclusion Criteria:

1. Known resistance or intolerance to ziprasidone
2. Medical contraindication to ziprasidone
3. Individuals on ziprasidone immediately prior to study enrollment
4. Prior or current treatment with clozapine
5. Diagnosis of eating disorder
6. Individuals whose sub-optimal adherence is related to inability to pay for BD medication treatment or inability to arrange transportation to BD treatment clinical visits
7. Concurrent medical condition or psychiatric illness, which in the opinion of the research psychiatrist, would interfere with the patient's ability to participate in the trial
8. Current substance dependence
9. High risk of harm to self or others
10. Female who is currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, M.D., Principal Investigator — Case Western Reserve University School of Medicine
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Medication Adherence Bipolar Disorder: Drug: Ziprasidone. Dosages were titrated for each participant up to a maximum of 160 mg/day from a minimum of 20 mg/day. Dosages were in pill form once per day.
  There was only one group for this study.
Period: Overall Study
Arm/Group | Medication Adherence Bipolar Disorder
Started | 30
Completed | 20
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Medication Adherence Bipolar Disorder
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (10.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Treatment Non-adherence Percentage as Measured by the Tablet Routines Questionnaire (TRQ)
Description: Scale Range: 0-100%. The score represents percentage of time that required medication doses were missed. Higher scores indicate lower medication adherence.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: Percentage of doses
Arm/Group | Medication Adherence Bipolar Disorder
Number analyzed (Participants) | 20
Percentage of doses
  Past week | 16.11 (16.46)
  Past month | 13.88 (14.08)

2. Secondary Outcome: Treatment Adherence Score as Measured by the Morisky Rating Scale
Description: Four item inventory taken by participant with Scale Range: 0-4. Lower scores indicate improved outcomes.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication Adherence Bipolar Disorder
Number analyzed (Participants) | 20
units on a scale | 2.90 (1.25)

3. Secondary Outcome: Attitude Toward Medication Score as Measured by the Drug Attitude Inventory
Description: Ten item inventory taken by the participant with a Scale Range: 0-10. Higher scores indicate improved outcomes.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication Adherence Bipolar Disorder
Number analyzed (Participants) | 20
units on a scale | 6.10 (3.08)

4. Secondary Outcome: Global Psychopathology Score as Measured by Clinical Global Impressions
Description: Global psychopathology will be measured with the Clinical Global Impressions (CGI) (Guy 1976) a widely used scale which evaluates illness severity on a 1 to 7 point continuum. Severity of illness ratings on the CGI have reported reliability scores ranging from 0.41-0.66 (Guy 1976). Lower scores indicate improved outcomes.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication Adherence Bipolar Disorder
Number analyzed (Participants) | 20
units on a scale | 2.25 (1.29)

5. Secondary Outcome: Social and Occupational Functioning Scale
Description: Life and Work Functional status will be evaluated using the Social and Occupational Functioning Scale (SOFAS), which is derived from the GAF (Global Assessment of Functioning). The GAF is a 100-point single-item scale which measures global functioning of psychiatric patients and is widely utilized in clinical studies involving Seriously Mentally Ill patients (Jones 1995). The reliability of the GAF ranges from 0.62-0.82. Higher scores indicate improved outcomes.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication Adherence Bipolar Disorder
Number analyzed (Participants) | 20
units on a scale | 54.40 (9.46)

6. Secondary Outcome: Montgomery Asberg Depression Rating Scale
Description: Scale Range: 0-60. Lower scores indicate better outcomes.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication Adherence Bipolar Disorder
Number analyzed (Participants) | 20
units on a scale | 12.35 (11.21)

7. Secondary Outcome: Young Mania Rating Scale
Description: Scale Range: 0-60. Lower scores indicate better outcomes.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication Adherence Bipolar Disorder
Number analyzed (Participants) | 20
units on a scale | 5.30 (5.82)

8. Secondary Outcome: Body Weight
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Medication Adherence Bipolar Disorder
Number analyzed (Participants) | 20
lbs | 210.75 (60.94)

9. Secondary Outcome: Quality of Life Score as Measured by 12-item Short Form Health Survey
Description: Scale Range: 1-99th percentile score. Higher scores indicate better outcomes.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication Adherence Bipolar Disorder
Number analyzed (Participants) | 20
units on a scale
  Norm-Based Standardized PCS Score | 41.13 (12.71)
  Norm-Based Standardized MCS Score | 42.00 (13.44)

ADVERSE EVENTS:
Arm/Group | Medication Adherence Bipolar Disorder
Serious Adverse Events (participants affected / at risk) | 12/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication Adherence Bipolar Disorder (N=30)
Rashes (Skin and subcutaneous tissue disorders) | 1 (1)
Psychiatric Hospitalization (Psychiatric disorders) | 5 (5)
High Blood Glucose (Metabolism and nutrition disorders) | 1 (2)
Swollen Tongue and Facial Distortion (General disorders) | 1 (1)
Car Accident (General disorders) | 1 (1) — Participant passed out while driving. The accident may have been related to new-onset elevated blood pressure.
Fall (General disorders) | 1 (1) — Participant fell down stairs while carrying dishes. Hospitalized with internal bleeding and a ruptured spleen.
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gallstones (Hepatobiliary disorders) | 1 (1) — Participant reported having had recurrent abdominal pain for many years. Sought treatment in December 2011 and was found to have gallstones.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No